CLINICAL TRIAL: NCT02553161
Title: Mechanism of Antidepressant-Related Dysfunctional Arousal in High-Risk Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Melissa Delbello, Principal Investigator, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DelBello/Singh AIM; R01MH105469 (NIH)
Record Dates: First submitted 2015-09-10; First posted 2015-09-17 (Estimated); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Depression; Anxiety; Bipolar Disorder
Keywords: Depression
MeSH Terms: conditions — Depression; Anxiety Disorders; Bipolar Disorder | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MED - Escitalopram with psychotherapy (Experimental): Youth will also be assigned a board certified child psychiatrist (Drs. Singh or Chang at Stanford; Drs. DelBello or Patino at UC), who will be blind to treatment condition and see youth weekly for the first 4 weeks, then biweekly until 16 weeks. Youth in the MED condition will be given the USFDA (US Food & Drug Administration) approved antidepressant, escitalopram for the treatment of depression or anxiety in youth and follow a standard dose titration schedule of 5 mg/day for 1 week, 10mg/day for 1 week, then with a target dose of 20-30 mg/day by 4 weeks.
  Interventions: Drug: Escitalopram
- No MED -Psychotherapy (Placebo Comparator): All participants (No MED and MED) will be assigned a study-trained therapist who will provide hour-long weekly individual cognitive behavioral psychotherapy (CBT) based on current evidence-based practices for the treatment of anxiety and depressive symptoms for youth.
  Interventions: Behavioral: Cognitive behavioral Psychotherapy
- Healthy Control (No Intervention): 60 (30 at Stanford, 30 at University of Cincinnati) 12- to 17-year old male and female typically developing healthy controls. Healthy controls will receive behavioral, neural, and physiological assessments at baseline only. healthy controls will be scanned at baseline only and serve as a reference group to determine whether MRI changes observed in the high-risk group from baseline to week 4 are toward or away from normal.

INTERVENTIONS:
Drug: Escitalopram — Youth in the MED condition will be given the USFDA approved antidepressant, escitalopram for the treatment of depression or anxiety in youth and follow a standard dose titration schedule of 5 mg/day for 1 week, 10mg/day for 1 week, then with a target dose of 20-30 mg/day by 4 weeks. Titration will be no faster than 5mg/week. This titration guideline was drawn from the escitalopram package insert for pediatric dosing, which states that target doses may be achieved by 4 weeks.
  Other Names: Lexapro
  Arms: MED - Escitalopram with psychotherapy
Behavioral: Cognitive behavioral Psychotherapy — All participants (No MED and MED) will be assigned a study-trained therapist who will provide hour-long weekly individual cognitive behavioral psychotherapy (CBT) based on current evidence-based practices for the treatment of anxiety and depressive symptoms for youth.
  Other Names: CBT
  Arms: No MED -Psychotherapy

SUMMARY:
A 16-week double blind, placebo-controlled investigation of escitalopram in adolescents with depression and/or anxiety with a family history of Bipolar Disorder. Subjects will be evaluated using semi-structured diagnostic interviews and symptom ratings, participate in a MRI scan and then randomized to treatment. Following randomization, high-risk youth will have visits every week for the first 4 weeks of treatment then biweekly up to 16 weeks during which time tolerability and ratings will be performed. MRI scan will be repeated at week 4.

DETAILED DESCRIPTION:
The primary goals of this proposal are to investigate the etiological mechanisms associated with antidepressant-related dysfunctional emotional arousal and to characterize baseline neurobiological risk factors that predict the development of dysfunctional emotional arousal in treatment seeking youth with a family history of BD.

Antidepressants have moderate benefit for treating mood and anxiety disorders in childhood but their effects on the developing brain are largely unknown. Antidepressants are among the most commonly prescribed medications used by youth in the United States and are used to treat many psychiatric disorders including depression, dysthymia and anxiety. However, recent reviews suggest that antidepressants provide only mild to moderate benefit. Moreover, a growing number of case reports and clinical studies have described antidepressant-related psychiatric adverse events such as aggression, psychosis, agitation, suicidal ideation, hypomania or mania, all behaviors associated with increased emotional arousal. Importantly, these adverse events are more likely to occur in children than adults. With younger ages of treatment combined with increased and repeated exposure during critical sensitive periods of neurodevelopment, these adverse events are becoming a rising concern for youth, and may lead to the development of serious psychopathologies in youth that carry an enormous burden of illness, such as bipolar disorder (BD). Given that BD typically begins before 18 years of age and with a depressive episode, there are millions of youth in the U.S. each year who experience their first bipolar episode as a depressive episode that is routinely treated with antidepressants. However, the mechanisms and risk factors through which antidepressants increase risk for developing adverse outcomes are largely unknown.

Youth with a family history of BD have a high likelihood of developing adverse responses to antidepressants, possibly because such youth are already vulnerable to developing dysfunctional emotional arousal and may use antidepressants to treat mood and anxiety symptoms. Indeed, a family history of BD is among the strongest risk factors for developing disorders of emotional arousal in youth. Twin and family studies have provided compelling evidence that having a parent with BD is associated with dramatic increases in risk for the offspring's development of disorders of emotional arousal compared with the general population. Moreover, when these offspring develop dysfunctional emotional arousal, their risk of developing BD increases even further. Antidepressants are commonly used to treat initial mood presentations; however, they may also accelerate the onset of dysfunctional emotional arousal in these high-risk youth. In this context, it becomes difficult to disentangle a natural illness progression from an antidepressant-related dysfunction leading to BD. Thus, there is a significant clinical dilemma regarding whether antidepressants should be prescribed to treat youth with a family history of BD, who also have DSM-5 (Diagnostic and Statistical Manual of Mental Disorders) depressive and anxiety disorders.

ELIGIBILITY:
Inclusion Criteria:

Inclusion - High-Risk Youth:

1. age 12 years, 0 mos. - 17 years, 11 mos.;
2. at least one parent or step-parent/guardian with whom the subject lives is willing to participate in research sessions;
3. the child and relative(s) are able and willing to give written informed assent/consent to participate, respectively;
4. the youth meets criteria for high-risk:

   * has at least one first degree relative with Bipolar I Disorder, as assessed by the Structured Clinical Interview for DSM (SCID; First et al. 1995), the Kiddie Schedule for Affective Disorders and Schizophrenia (KSADS-PL, Kaufman et al., 1997), and the Family History-Research Diagnostic Criteria (FH-RDC; Andreasen et al., 1977);
   * the youth shows evidence of current significant depressive or anxiety symptoms as determined by a current Childhood Depression Rating Scale-Revised (CDRS-R, Poznanski et al.,1984) score > 35 and/or a current Pediatric Anxiety Rating Scale (PARS, 2002) score > 15.

Inclusion - Healthy Controls:

1. age 12 years, 0 mos. - 17 years, 11 mos.;
2. at least one parent or step-parent/guardian with whom the subject lives is willing to participate in research sessions;
3. the child and relative(s) are able and willing to give written informed assent/consent to participate, respectively;
4. no personal or family history of any psychopathology as assessed by the KSADS-PL structured clinical interview (Kaufman et al., 1997) and the Family History-Research Diagnostic Criteria (FH-RDC; Andreasen et al., 1977).

Exclusion Criteria:

Exclusion - High-Risk Youth & Healthy Controls:

1. any history of syndromal bipolar I or II disorder (i.e., history of mania, mixed episode, or major depression with hypomania);
2. a history of previous antidepressant exposure
3. a DSM-5 diagnosis of autism, pervasive developmental disorder, OCD(Obsessive-Compulsive Disorder), PTSD, Tourette's disorder, or any psychotic disorder including schizophrenia;
4. evidence of mental retardation (IQ < 70) as determined by the Weschler Abbreviated Scale of Intelligence (WASI; Psychological Corporation, 1999);
5. comorbid neurologic diseases such as seizure disorder;
6. Drug or alcohol abuse or dependence disorders in the 4 months prior to study recruitment, although a lifetime history of substance or alcohol disorders can be present if the child has been abstinent for at least 6 months (see further discussion below);
7. evidence of an unstable medical or psychiatric disorder that requires immediate hospitalization or other emergency medical treatment;
8. a positive pregnancy test; participants will be encouraged but not mandated to discuss a positive pregnancy test with their guardians and we will follow local laws.
9. any contraindication for MRI, including metal in the body related to an injury or surgery (e.g., surgical clips, metal fragments in the eyes), piercings that cannot be removed, braces, or permanent retainers.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 214 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2022-07 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Baseline-endpoint change in prefrontal-amygdala functional connectivity by Scan. | Baseline to 16 weeks
  Study the neural mechanisms of antidepressant-related dysfunctional arousal by ensuring that the treatment assignment precedes the 4-week scan, and the 4-week scan precedes the assessment of highest arousal measured between 4 and 16 weeks.The change in amygdala hyperactivity from the baseline to 4-week scan will be treated as the outcome and the treatment status (MED vs. No MED) will be treated as the predictor variable. The primary outcome is the level of post-treatment arousal (highest after the 4-week scan). The early change (baseline to 4 weeks) in amygdala hyperactivity, treatment assignment (MED vs. No MED), and the interaction between the two will be the predictors of arousal.

SECONDARY OUTCOMES:
Week 4- endpoint change in mood by and arousal ratings | Between week 4 and 16
  We will also explore subgroups of arousal due to worsening symptom severities of mania, anxiety, depression, psychosis, suicidality, and anxiety, using clinical, self, and parent (e.g. TEASAP) report measures of emotional reactivity and lability, and reaction times during the Continuous Performance Task with Emotional and Neutral Distracters (CPT-END) as secondary predictors of dysfunctional emotional arousal.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa P DelBello, MD, MS, Principal Investigator — University of Cincinnati; Manpreet K Singh, MD,MS, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford University, Stanford, California
  - University of Cincinnati, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Honeycutt DC, Blom TJ, Ramsey LB, Strawn JR, Bruns KM, Welge JA, Patino LR, Singh MK, DelBello MP. Pharmacogenetic Factors Influence Escitalopram Pharmacokinetics and Adverse Events in Youth with a Family History of Bipolar Disorder: A Preliminary Study. J Child Adolesc Psychopharmacol. 2024 Feb;34(1):42-51. doi: 10.1089/cap.2023.0073. PMID 38377518